CLINICAL TRIAL: NCT05430867
Title: Efficacy and Safety of Memantine and Sodium Oligomannate in Patients With Moderate to Severe Alzheimer's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2022LSK-042
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-06

CONDITIONS: Treatment; Efficacy; Safety; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine; GV-971

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Memantine monotherapy group (Experimental): Memantine 20mg once-daily
  Interventions: Drug: Memantine Oral Tablet
- GV-971 monotherapy group (Experimental): GV-971 450mg twice a day
  Interventions: Drug: GV-971 capsule
- Memantine combined with GV-971 group (Experimental): Memantine 20mg once-daily plus GV-971 450mg twice a day
  Interventions: Drug: Memantine Oral Tablet; Drug: GV-971 capsule

INTERVENTIONS:
Drug: Memantine Oral Tablet — Memantine 20mg once-daily
  Other Names: Memantine
  Arms: Memantine combined with GV-971 group; Memantine monotherapy group
Drug: GV-971 capsule — GV-971 450mg twice a day
  Other Names: GV-971
  Arms: GV-971 monotherapy group; Memantine combined with GV-971 group

SUMMARY:
Alzheimer's disease (AD) is the main cause of dementia. At present, AD is incurable. Memantine is recommended for the treatment of moderate and severe AD patients. Sodium oligomannate (GV-971) is a marine-derived oligosaccharide. It is proposed that it can reconstitute the gut microbiota, and inhibit neuroinflammation in the brain as observed in animal models. It reduces Aβ deposition in the brain of Aβ-transgenic mice. The reduction in both Aβ deposition and neuroinflammation may synergistically contribute to the improvement of cognitive impairment and delay the progress of the disease. China Food and Drug Administration（CFDA）approved it for the treatment of mild to moderate AD in 2019. Due to the different mechanism of memantine and GV-971, theoretically, they may synergistically improve cognitive function and delay disease progression. However, there is a lack of data on their effectiveness and safety. Therefore, the purpose of this study is to compare the efficacy and safety of memantine and GV-971 monotherapy and combination therapy in patients with moderate to severe AD, which is of great significance for guiding the treatment of moderate and severe AD.

ELIGIBILITY:
Inclusion Criteria:

* age of 50-80 years old , either sex;
* met the diagnostic criteria for suspected AD;
* moderate to severe AD patients(5 points ≤Mini-Mental State Examination total score≤14 points);
* total Hachinski ischemic scale (HIS) score ≤4 points;
* memory loss for at least 12 months, with a progressive deterioration;
* brain MRI scan suggesting a significant possibility of AD;
* no obvious physical signs during nervous system examination;
* stable and reliable caregivers;
* elementary school or higher education level;
* signed an informed consent form.

Exclusion Criteria:

* previous nervous system diseases ;
* mental illness;
* unstable or severe heart, lung, liver, kidney, or hematopoietic diseases;
* uncorrectable visual and auditory disorders;
* simultaneous use of cholinesterase inhibitors, memantine or GV-971.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
cognitive function | baseline, week 12, week 24, week 36,week 48
  the change of Severe Impairment Battery score （The total score ranges from 0 to 100，higher scores mean a better outcome）from baseline at week 48